CLINICAL TRIAL: NCT02787863
Title: Pathogenetic Justification and Clinical and Immunological Efficiency of Application Bacterial Vaccines at Adult Patients With Bronchopulmonary Pathology
Brief Title: Clinical and Immunological Efficiency of Bacterial Vaccines at Adult Patients With Bronchopulmonary Pathology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mikhael Petrovich Kostinov (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Mikhael Petrovich Kostinov, MD, PhD, Chief of Laboratory of Vaccines and Allergotherapy of allergic diseases, Russian Academy of Medical Sciences
Organization: Russian Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115030370013
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Pneumococcal Infections
Keywords: Pneumococcal vaccines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- COPD with Prevenar-13 (1) (Experimental): 33 patients with COPD. Standard therapy with Prevenar-13.
  Interventions: Biological: Prevenar-13
- Asthma with Prevenar 13 (2) (Experimental): 34 patients with asthma. Standard therapy with Prevenar 13.
  Interventions: Biological: Prevenar-13
- COPD with Pneumo-23 (3) (Experimental): 25 patients with COPD. Standard therapy with Pneumo-23.
  Interventions: Biological: Pneumo-23
- Asthma with Pneumo-23 (4) (Experimental): 25 patients with asthma. Standard therapy with Pneumo-23.
  Interventions: Biological: Pneumo-23
- COPD with Pneumo-23/Prevenar-13 (5) (Experimental): 32 patients with COPD. Standard therapy, vaccinated with pneumococcal polysaccharide vaccine/pneumococcal conjugate vaccine (PPV23/PCV13).
  Interventions: Biological: Prevenar-13; Biological: Pneumo-23
- Asthma with Pneumo-23/Prevenar-13 (6) (Experimental): 18 patients with Asthma. Standard therapy, vaccinated with PPV23/PCV13.
  Interventions: Biological: Prevenar-13; Biological: Pneumo-23
- COPD with Prevenar-13/Pneumo-23 (7) (Experimental): 25 patients with COPD. Standard therapy, vaccinated with PCV13/PPV23.
  Interventions: Biological: Prevenar-13; Biological: Pneumo-23
- Asthma with Prevenar-13/Pneumo-23 (8) (Experimental): 27 patients with Asthma. Standard therapy, vaccinated with PCV13/PPV23.
  Interventions: Biological: Prevenar-13; Biological: Pneumo-23

INTERVENTIONS:
Biological: Prevenar-13 — Conjugate 13 serotype pneumococcal vaccine
  Other Names: PCV13
  Arms: Asthma with Pneumo-23/Prevenar-13 (6); Asthma with Prevenar 13 (2); Asthma with Prevenar-13/Pneumo-23 (8); COPD with Pneumo-23/Prevenar-13 (5); COPD with Prevenar-13 (1); COPD with Prevenar-13/Pneumo-23 (7)
Biological: Pneumo-23 — Polysaccharide 23-valent pneumococcal vaccine.
  Other Names: PPV23
  Arms: Asthma with Pneumo-23 (4); Asthma with Pneumo-23/Prevenar-13 (6); Asthma with Prevenar-13/Pneumo-23 (8); COPD with Pneumo-23 (3); COPD with Pneumo-23/Prevenar-13 (5); COPD with Prevenar-13/Pneumo-23 (7)

SUMMARY:
Goal: to to examine the formation of postvaccination immunity and evaluate the therapeutic effect of bacterial vaccines in patients with inflammation diseases of bronchopulmonary system. Objectives of the study: assessment of microbiocenosis mucous membranes of the upper respiratory tract in patients with bronchopulmonary pathology before and after use of bacterial vaccines. Identification of mayor lymphocytes subpopulations in patients in the dynamics of the vaccination process. Study the profile of humoral immune response in patients under different schemes of vaccination. Assessment of the clinic and functional status bronchopulmonary system in the immunized patients.

DETAILED DESCRIPTION:
Methods:

1. Immunoglobulin G (IgG)-antibodies against Streptococcus pneumoniae (S. pneumoniae) - solid-phase enzyme-linked immunoelectrodiffusion essay (ELISA).
2. General levels of Immunoglobulin A (IgA), Immunoglobulin M (IgM), IgG, Immunoglobulin E (IgE) in sera - radial immunodiffusion.
3. Phagocytic activity (granulocytes, monocytes), nitroblue tetrazolium test; T-lymphocytes, T-helpers (cluster of differentiation, CD3+CD4+), cytotoxic T-lymphocytes (СD3+CD8+), B-lymphocytes (CD19+); NK-cells (CD3-CD16+CD56+), NKT-cells (CD3+CD16+CD56+), activated T-cells (human leucocyte antigens, CD3+HLA DR+), CD3-HLA DR+.
4. Microbiological examination of sputum.
5. Determining the clinical effectiveness of vaccination.

   * the number of exacerbations of chronic bronchopulmonary pathology for the year prior to vaccination and during the first and fourth years after vaccination;
   * the number of courses of antibiotic therapy a year prior to vaccination and during the first and fourth years after immunization;
   * the number of hospitalizations for acute exacerbations of chronic bronchopulmonary disease during the year prior to vaccination and during the first and fourth years after immunization.
6. Method of estimating quality of life associated with health in patients with chronic bronchopulmonary pathology (asthma control questionnaire (ACQ-5), COPD assessment test (CAT)).

Characteristics of variables (arms 1-8).

1. The age of patients (years): mean (standard deviation) [min; median; max] for normally distributed variables; median [Q25; Q75] - for variables with distribution different from normal.
2. Gender: male/female.
3. Indicators of immune status

   * IgG antibodies to S. pneumoniae
   * IgA, g/l [0,4-3,5]
   * IgM, g/l [0,7-2,8]
   * IgG, g/l [8-18]
   * IgE, IU/ml [< 100]
   * Phagocytic index (granulocyte), % [82-90]
   * Phagocytic index (monocytes), % [75-85]
   * The participation rate of spontaneous NBT-test (neutrophils), % with intensity of 0.2.e. [7-14]
   * The index of activity induced NBT-test (neutrophils), % if intensity >of 0.36.e. [>28]
   * The percentage of NBT-positive cells in spontaneous test, % [2-19]
   * Circulating immune complexes (CEC) cond. units [0,055-0,11]
   * CD3+, % [55-80]
   * CD3+CD4+, % [31-49]
   * CD3+CD8+, % [12-30]
   * CD19+, % [5-19]
   * CD3-CD16+CD56+, % [6-20]
   * CD3+CD16+CD56+, % [<10]
   * CD3-HLA DR+, % [5-20]
   * CD3+HLA DR+, % [<12]
   * CD45RO. The reference value = 0,2.
4. Microbiological examination of sputum: frequency of selection of certain microorganisms are presented as absolute number of cases and % in the respective groups.
5. Evaluation of early post-vaccination period

   * The General condition (satisfactory/unsatisfactory)
   * Local reactions: pain (n/%), redness (n/%, cm), consolidation (n/%, cm)
   * General reactions:

     * Temperature 37,0-37,5 (n/%)
     * Temperature of 37.6-38,5 (n/%)
     * A temperature of 38.6 and > (n/%)
     * Headache (n/%)
     * Malaise, fatigue (n/%)
     * Joint pain (n/%)
     * Muscle pain (n/%)
6. Health related quality of life (HRQoL): CAT-test (for Chronic obstructive pulmonary disease (COPD) patients), ACQ-5 (for asthma patients).

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes from 18 years with a diagnosis of COPD or Bronchial Asthma;
* The presence of signed and dated informed consent to participate in a clinical study;
* The ability to perform the requirements of the Protocol;
* For women of childbearing age is a negative result of a pregnancy test before vaccination.

Diagnostic criteria for:

- COPD: dyspnea: progressive (worsens over time), increases with exertion, persistent; chronic cough (may appear sporadically and may be unproductive); chronic expectoration; the impact of risk factors in the medical history (Smoking, occupational dust pollutants and chemicals); widespread wheeze on auscultation of the chest and/or distant wheezing in the chest; family history of COPD; spirometric data confirming the presence of fixed bronchial obstruction.

Exclusion Criteria:

* Vaccination against pneumococcal infection in anamnesis;
* Application of preparations of immune globulin or blood transfusion within last three months prior to clinical studies;
* Prolonged use (more than 14 days) immunosuppressants or other immunosuppressive drugs within 6 months prior to the start of the study;
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including Human Immunodeficiency Virus (HIV) infection;
* A history or currently hematologic and other cancers;
* A positive reaction for HIV infection, viral hepatitis B and hepatitis C;
* The presence of respiratory, cardio-vascular insufficiency, impaired liver and kidney function, established during a physical examination at visit number 1;
* Pronounced congenital defects or serious chronic diseases in the acute stage, including any clinically important exacerbation of chronic diseases of the liver, kidney, cardiovascular, nervous system, mental diseases or metabolic disorders, confirmed by the history or objective examination (pulmonary: cystic fibrosis, lung abscess, empyema, active tuberculosis; extra-pulmonary: congestive heart failure, malabsorption, chronic renal and hepatic failure, cirrhosis, malignancy, immunodeficiency, cirrhosis of the liver);
* Severe allergic reactions in anamnesis, autoimmune disease;
* The presence of acute infectious and/or communicable illnesses within 1 month prior to study;
* History of chronic alcohol abuse and/or drug use;
* Exacerbation of chronic diseases;
* Breastfeeding;
* Pregnancy;
* Participation in any other clinical study within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei D Protasov, Professor, Principal Investigator — Samara State Medical University; Mikhael P Kostinov, Professor, Principal Investigator — Institute of Sera and Vaccines RAS, Moscow; Mikhael P Kostinov, Professor, Study Chair — Institute of Sera and Vaccines RAS, Moscow; Aleksander V Zhestkov, Professor, Study Chair — Samara State Medical University
Locations (2):
- Russia (2):
  - Samara State Medical Univercity, Samara, Samara Oblast
  - Institute of Sera and Vaccines RAS, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Protasov AD. Pneumococcal vaccination in patients with chronic broncho-pulmonary disease (literature review). The Bulletin of Contemporary Clinical Medicine. 6(2): 60-65, 2013.
- [Result] Protasov AD, Zhestkov AV, Kostinov MP. First results of 13-valent pneumococcal conjugate vaccine treatment in patients with chronic bronchopulmonary diseases: evaluation safety and tolerability. Russian Allergology Journal 4: 18-23, 2013.
- [Result] Protasov AD.COMPARATIVE EVALUATION OF THE EFFECTIVENESS OF PNEUMOCOCCAL VACCINATION WITH 13-VALENT CONJUGATE AND 23-VALENT POLYSACCHARIDE VACCINE IN PATIENTS WITH COPD. Russian Allergology Journal 4: 12-17, 2014.
- [Result] Kostinov MP, Protasov AD, Zhestkov AV, Polishuk VB. Promising data with pneumococcal 13-valent conjugate vaccine in adult patients with chronic bronchopulmonary pathology. Pulmonology 4: 57-63, 2014
- [Result] Protasov AD. Comparative evaluation of the effectiveness of vaccination against pneumococcal infection in patients with bronchial asthma with the use of 13-valent conjugate and 23-valent polysaccharide vaccine. Pulmonology. 5: 52-56, 2014
- [Result] Kostinov MP, Zhestkov AV, Protasov AD, Kostinova TA, Pakhomov DV, Chebykina AV, Magarshak OO.Comparative analysis of dynamics of indicators of quality of life in patients with chronic obstructive pulmonary disease on the background of vaccination against pneumococcal disease using the 13-valent conjugate and 23-valent polysaccharide vaccine. Pulmonology 25(2): 163-166, 2015
- [Result] Protasov AD, Kostinov MP, Zhestkov AV, Shteiner ML, Magarshak OO, Kostinova TA, Ryzhov AA, Pakhomov DV, Blagovidov DA, Panina MI. [Choice of optimal vaccination tactics against pneumococcal infection from immunological and clinical standpoints in patients with chronic obstructive pulmonary disease]. Ter Arkh. 2016;88(5):62-69. doi: 10.17116/terarkh201688562-69. Russian. PMID 27239929
- [Result] Protasov AD, Zhestkov AV, Kostinov MP, Shteiner ML, Tezikov YV, Lipatov IS, Yastrebova NE, Kostinova AM, Ryzhov AA, Polishchuk VB. [Analysis of the effectiveness and long-term results of formation of adaptive immunity in the use of various medications and vaccination schemes against pneumococcal infection in patients with chronic obstructive pulmonary disease]. Ter Arkh. 2017;89(12. Vyp. 2):165-174. doi: 10.17116/terarkh20178912165-174. Russian. PMID 29488477
- [Result] Protasov AD, Zhestkov AV, Kostinov MP, Korymasov EA, Shteyner ML, Tezikov YV, Lipatov IS, Reshetnikova VP, Lavrent'yeva NE. Long-term clinical efficacy and a possible mechanism of action of different modes of pneumococcal vaccination in asthma patients. Pulmonology 28(2): 193-199, 2018.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB approval - 05 SEP 2012 (protocol #122, Samara State Medical University). Dates of recruitment period - 06 SEP 2012 - 07 JUL 2013. FPFV - 06 SEP 2012. LPLV - 07 JUL 2017. Types of location - Samara State Medical University, Institute of Sera and Vaccines RAS (Russian Federation).
Pre-assignment Details: 219 patients were examined and monitored for 4 years. Distributed in a row, first to the PCV13 group, then to the PPV23, PPV23/PCV13 and PCV13/PPV23 groups for COPD and asthma.
Groups:
- COPD - Prevenar-13 (1): 33 patients with COPD. Prevenar-13 (PCV13) vaccination.
- Asthma - Prevenar-13 (2): 34 patients with asthma. Prevenar-13 (PCV13) vaccination.
- COPD - Pneumo-23 (3): 25 patients with COPD. Pneumo-23 (PPV23) vaccination.
- Asthma - Pneumo-23 (4): 25 patients with asthma. Pneumo-23 (PPV23) vaccination.
- COPD - Pneumo-23/Prevenar-13 (5): 32 patients with COPD, PPV23/PCV13.
  PPV23 vaccination was first, PCV13 vaccination was after 12 months after PPV23.
- Asthma - Pneumo-23/Prevenar-13 (6): 18 patients with Asthma. PPV23/PCV13.
  PPV23 vaccination was first, PCV13 vaccination was after 12 months after PPV23.
- COPD - Prevenar-13/Pneumo-23 (7): 25 patients with COPD. PCV13/PPV23 vaccination.
  PCV13 vaccination was first, PPV23 vaccination was after 2 months after PCV13.
- Asthma - Prevenar-13/Pneumo-23 (8): 27 patients with Asthma. PCV13/PPV23 vaccination.
  PCV13 vaccination was first, PPV23 vaccination was after 2 months after PCV13.
Period: Overall Study
Arm/Group | COPD - Prevenar-13 (1) | Asthma - Prevenar-13 (2) | COPD - Pneumo-23 (3) | Asthma - Pneumo-23 (4) | COPD - Pneumo-23/Prevenar-13 (5) | Asthma - Pneumo-23/Prevenar-13 (6) | COPD - Prevenar-13/Pneumo-23 (7) | Asthma - Prevenar-13/Pneumo-23 (8)
Started | 33 | 34 | 25 | 25 | 32 | 18 | 25 | 27
1 Year After Vaccination | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
4 Years After Vaccination | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
Completed | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
Not Completed | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- COPD With Pneumo-23/Prevenar-13 (5): 32 patients with COPD. Standard therapy, vaccinated with PPV23/PCV13.
  Prevenar-13: Conjugate 13 serotype pneumococcal vaccine
  Pneumo-23: Polysaccharide 23-valent pneumococcal vaccine.
- Total: Total of all reporting groups
Arm/Group | COPD With Prevenar-13 (1) | Asthma With Prevenar 13 (2) | COPD With Pneumo-23 (3) | Asthma With Pneumo-23 (4) | COPD With Pneumo-23/Prevenar-13 (5) | Asthma With Pneumo-23/Prevenar-13 (6) | COPD With Prevenar-13/Pneumo-23 (7) | Asthma With Prevenar-13/Pneumo-23 (8) | Total
Number analyzed (Participants) | 33 | 34 | 25 | 25 | 32 | 18 | 25 | 27 | 219
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 patients died of chronic pulmonary hypertension, 2 patients withdrawal of informed consent during 1-st year of the trial (1 subject of I group, I subject of II group, 2 subjects of III group).
  Participants
    number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27 | 215
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 17 | 25 | 12 | 23 | 18 | 16 | 15 | 22 | 148
    >=65 years | 15 | 8 | 11 | 2 | 14 | 2 | 10 | 5 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: 2 patients died of chronic pulmonary hypertension, 2 patients withdrawal of informed consent during 1-st year of the trial (1 subject of I group, I subject of II group, 2 subjects of III group).
  years
    number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27 | 215
    (all) | 63.6 (8.7) | 52.5 (15.3) | 59 (12.4) | 49.1 (13.3) | 63.9 (10.9) | 48.5 (14.3) | 60.5 (12.1) | 49.3 (15.4) | 56.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: 2 patients died of chronic pulmonary hypertension, 2 patients withdrawal of informed consent during 1-st year of the trial (1 subject of I group, I subject of II group, 2 subjects of III group).
  Participants
    number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27 | 215
    Female | 11 | 22 | 10 | 19 | 13 | 12 | 7 | 18 | 112
    Male | 21 | 11 | 13 | 6 | 19 | 6 | 18 | 9 | 103
Region of Enrollment [Number; unit: participants]
  Russia | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27 | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Without Exacerbations of the Underlying Disease, Antibiotic Use and Hospitalisation.
Description: Number of patients without exacerbations of the underlying disease, antibiotic use and hospitalisation.
Time Frame: Baseline (1 year prior to vaccination), 1 year after vaccination, 4 years after vaccination
Measure: Count of Participants; unit: Participants
Groups:
- COPD - Prevenar-13 (1): 32 patients with COPD. Prevenar-13 (PCV13) vaccination.
- Asthma - Prevenar-13 (2): 33 patients with asthma. Prevenar-13 (PCV13) vaccination.
- COPD - Pneumo-23 (3): 23 patients with COPD. Pneumo-23 (PPV23) vaccination.
Arm/Group | COPD - Prevenar-13 (1) | Asthma - Prevenar-13 (2) | COPD - Pneumo-23 (3) | Asthma - Pneumo-23 (4) | COPD - Pneumo-23/Prevenar-13 (5) | Asthma - Pneumo-23/Prevenar-13 (6) | COPD - Prevenar-13/Pneumo-23 (7) | Asthma - Prevenar-13/Pneumo-23 (8)
Number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
Participants
  Without exacerbations, 1 year prior to vaccination | 3 | 5 | 1 | 0 | 3 | 1 | 1 | 2
  Without exacerbations, 1 year after vaccination | 22 | 28 | 17 | 14 | 11 | 7 | 18 | 20
  Without exacerbations, 4 years after vaccination | 10 | 11 | 4 | 4 | 2 | 5 | 13 | 13
  Without antibiotics, 1 year prior to vaccination | 6 | 12 | 2 | 6 | 5 | 4 | 2 | 7
  Without antibiotics, 1 year after vaccination | 25 | 29 | 18 | 16 | 14 | 9 | 19 | 16
  Without antibiotics, 4 years after vaccination | 12 | 21 | 5 | 8 | 11 | 7 | 13 | 18
  Without hospitalisat, 1 year prior to vaccination | 13 | 18 | 10 | 15 | 15 | 11 | 9 | 20
  Without hospitalisat, 1 year after vaccination | 29 | 32 | 21 | 24 | 25 | 17 | 21 | 21
  Without hospitalisat, 4 years after vaccination | 24 | 27 | 13 | 16 | 21 | 14 | 23 | 26
Statistical Analysis 1: Comparison: COPD - Prevenar-13 (1) vs Asthma - Prevenar-13 (2) vs COPD - Pneumo-23 (3) vs Asthma - Pneumo-23 (4) vs COPD - Pneumo-23/Prevenar-13 (5) vs Asthma - Pneumo-23/Prevenar-13 (6) vs COPD - Prevenar-13/Pneumo-23 (7) vs Asthma - Prevenar-13/Pneumo-23 (8); Test type: Other; p < 0.05, McNemar

2. Primary Outcome: The Number of Exacerbations of the Underlying Disease, Antibiotic Use and Hospitalisation
Description: The number of exacerbations of the underlying disease, antibiotic use and hospitalisation. The average number of exacerbations per 1 patient = total exacerbations in the group / number of patients in the group. This is not a mean value.
Time Frame: Baseline (1 year prior to vaccination), 1 year after vaccination, 4 years after vaccination
Measure: Number; unit: Events per 1 patient
Groups:
- COPD - Prevenar-13 (9): 32 patients with COPD. Prevenar-13 (PCV13) vaccination.
- Asthma - Prevenar-13 (10): 33 patients with asthma. Prevenar-13 (PCV13) vaccination.
- COPD - Pneumo-23 (11): 23 patients with COPD. Pneumo-23 (PPV23) vaccination.
- Asthma - Pneumo-23 (12): 25 patients with asthma. Pneumo-23 (PPV23) vaccination.
- COPD - Pneumo-23/Prevenar-13 (13): 32 patients with COPD, PPV23/PCV13.
  PPV23 vaccination was first, PCV13 vaccination was after 12 months after PPV23.
- Asthma - Pneumo-23/Prevenar-13 (14): 18 patients with Asthma. PPV23/PCV13.
  PPV23 vaccination was first, PCV13 vaccination was after 12 months after PPV23.
- COPD - Prevenar-13/Pneumo-23 (15): 25 patients with COPD. PCV13/PPV23 vaccination.
  PCV13 vaccination was first, PPV23 vaccination was after 2 months after PCV13.
- Asthma - Prevenar-13/Pneumo-23 (16): 27 patients with Asthma. PCV13/PPV23 vaccination.
  PCV13 vaccination was first, PPV23 vaccination was after 2 months after PCV13.
Arm/Group | COPD - Prevenar-13 (9) | Asthma - Prevenar-13 (10) | COPD - Pneumo-23 (11) | Asthma - Pneumo-23 (12) | COPD - Pneumo-23/Prevenar-13 (13) | Asthma - Pneumo-23/Prevenar-13 (14) | COPD - Prevenar-13/Pneumo-23 (15) | Asthma - Prevenar-13/Pneumo-23 (16)
Number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
Events per 1 patient
  The number of exacerbations (before vaccination) | 1.97 | 2.24 | 2.13 | 2.68 | 2.22 | 2.39 | 2.52 | 1.89
  The number of exacerbations (1-st year) | 0.41 | 0.24 | 0.35 | 0.64 | 2.19 | 1.22 | 0.32 | 0.44
  The number of exacerbations (4-th year) | 1.16 | 0.85 | 1.52 | 1.2 | 1.72 | 1 | 0.84 | 0.56
  The number of antibiotic use (before vaccination) | 1.66 | 1.12 | 1.87 | 1.68 | 1.91 | 1.72 | 2.12 | 1.44
  The number of antibiotic use (1-st year)) | 0.31 | 0.12 | 0.3 | 0.56 | 1.59 | 1.06 | 0.24 | 0.48
  The number of antibiotic use (4-th year)) | 1.19 | 0.69 | 1.69 | 1.44 | 1 | 1.06 | 0.8 | 0.56
  The number of hospitalisation (before vaccination) | 0.88 | 0.73 | 0.87 | 0.56 | 0.94 | 0.56 | 0.84 | 0.48
  The number of hospitalisation (1-st year) | 0.13 | 0.03 | 0.09 | 0.04 | 0.47 | 0.06 | 0.16 | 0.26
  The number of hospitalisation (4-th year) | 0.63 | 0.3 | 0.96 | 0.56 | 0.47 | 0.44 | 0.2 | 0.04
Statistical Analysis 1: Comparison: COPD - Prevenar-13 (9) vs Asthma - Prevenar-13 (10) vs COPD - Pneumo-23 (11) vs Asthma - Pneumo-23 (12) vs COPD - Pneumo-23/Prevenar-13 (13) vs Asthma - Pneumo-23/Prevenar-13 (14) vs COPD - Prevenar-13/Pneumo-23 (15) vs Asthma - Prevenar-13/Pneumo-23 (16); Test type: Other; p < 0.05, McNemar

3. Secondary Outcome: Seeding Frequency S. Pneumoniae From Sputum in Patients With COPD
Description: Seeding frequency S. pneumoniae from sputum in patients with COPD
Time Frame: Baseline, after 1 and 4 years after vaccination
Measure: Number; unit: Number of Participants with S. Pneumonia
Arm/Group | COPD - Prevenar-13 (9) | Asthma - Prevenar-13 (10) | COPD - Pneumo-23 (11) | Asthma - Pneumo-23 (12) | COPD - Pneumo-23/Prevenar-13 (13) | Asthma - Pneumo-23/Prevenar-13 (14) | COPD - Prevenar-13/Pneumo-23 (15) | Asthma - Prevenar-13/Pneumo-23 (16)
Number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
Number of Participants with S. Pneumonia
  S. pneumoniae in sputum at baseline | 21 | 12 | 18 | 10 | 18 | 5 | 14 | 12
  S. pneumoniae in sputum after 1 year | 2 | 0 | 5 | 4 | 1 | 0 | 0 | 0
  S. pneumoniae in sputum after 4 years | 14 | 5 | 12 | 6 | 10 | 3 | 6 | 2

4. Secondary Outcome: Average CAT (COPD) and ACQ-5 (Asthma) Score
Description: CAT - COPD Assessment Test, min. = 0, max. = 40, higher scores mean a worse outcome.
  ACQ-5 - Asthma control questionnaire, min. = 0, max. = 6, higher scores mean a worse outcome.
Time Frame: Baseline, after 1 and 4 years after vaccination
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | COPD - Prevenar-13 (9) | Asthma - Prevenar-13 (10) | COPD - Pneumo-23 (11) | Asthma - Pneumo-23 (12) | COPD - Pneumo-23/Prevenar-13 (13) | Asthma - Pneumo-23/Prevenar-13 (14) | COPD - Prevenar-13/Pneumo-23 (15) | Asthma - Prevenar-13/Pneumo-23 (16)
Number analyzed (Participants) | 32 | 33 | 23 | 25 | 32 | 18 | 25 | 27
score on a scale
  Baseline | 21.8 [3 to 38] | 1.8 [0.6 to 2.2] | 22.8 [2 to 37] | 2 [1.4 to 2.2] | 16.8 [4 to 34] | 1.1 [0.5 to 2.2] | 23.4 [3 to 39] | 1.6 [0 to 3.6]
  1 year after vaccination | 11.5 [7 to 19.5] | 0.6 [0.2 to 1] | 14 [6.5 to 20] | 0.8 [0.4 to 2] | 11.5 [6 to 15.8] | 0.5 [0.2 to 1.1] | 11 [8 to 20] | 0.4 [0.2 to 0.9]
  4 years after vaccination | 18.2 [5 to 32] | 0.8 [0.4 to 1.4] | 20.5 [4 to 35] | 1.4 [1 to 1.8] | 15.1 [4 to 28] | 0.8 [0.4 to 1.35] | 19 [12 to 24] | 1 [0.5 to 1.2]

5. Secondary Outcome: Phagocytic Activity in Patients With COPD at Baseline, 1, 2, and 6 Weeks After PCV13 and PPV13 Vaccination
Description: Phagocytic index (granulocytes), phagocytic index (monocytes), activity of a spontaneous HCT test (neutrophils), activity of an induced HCT test (neutrophils), percentage of HCT-positive white blood cells in a spontaneous test. The phagocytic index was calculated according to the following formula: phagocytic index = (total number of engulfed cells/total number of counted macrophages) × (number of macrophages containing engulfed cells/total number of counted macrophages) × 100 (phagocytic index)
  The phagocytic index was calculated by counting at least 100 bacteria phagocytized by certain number of phagocytic cells/macrophages and expressed following formula (Mamnur Rashid 1997):
  Phagocytic index = Total no. of phagocytized bacteria /No of phagocytic cells phagocytizing bacteria.
  Activation index = % formazan positive cells (FPC) in NBT stimulated / % formazan positive cells (FPC) in NBT Spontaneous.
Time Frame: Baseline, 1, 2, 6 weeks after PCV13 and PPV13 vaccination
Population: Phagocytic index (granulocytes) - %, phagocytic index (monocytes) - %, activity of a spontaneous HCT test (neutrophils) - %, activity of an induced HCT test (neutrophils) - %, percentage of HCT-positive white blood cells in a spontaneous test - %.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COPD - Prevenar-13 (9) | COPD - Pneumo-23 (11)
Number analyzed (Participants) | 20 | 20
score on a scale
  Phagocytic index (granulocytes) - baseline | 65 (7.6) | 63 (5.5)
  Phagocytic index (granulocytes) - 1 week | 71 (8.2) | 65 (5.4)
  Phagocytic index (granulocytes) - 2 weeks | 84 (3.6) | 64.3 (4.8)
  Phagocytic index (granulocytes) - 6 weeks | 85 (3.2) | 66.5 (5.8)
  Phagocytic index (monocytes) - baseline | 72.1 (5.4) | 74.6 (5.2)
  Phagocytic index (monocytes) - 1 week | 74.1 (4.6) | 75.3 (5.7)
  Phagocytic index (monocytes) - 2 weeks | 74.4 (4.5) | 76.3 (4.1)
  Phagocytic index (monocytes) - 6 weeks | 77.3 (3.7) | 78.1 (6.6)
  activity of a spontaneous HCT test - baseline | 4 (1.3) | 5 (2.2)
  activity of a spontaneous HCT test - 1 week | 7.5 (3.1) | 5 (2.3)
  activity of a spontaneous HCT test - 2 weeks | 12.5 (4.7) | 7.2 (1.9)
  activity of a spontaneous HCT test - 6 weeks | 14.1 (4.4) | 6.9 (1.8)
  activity of an induced HCT test - baseline | 11 (3.4) | 9.3 (2.6)
  activity of an induced HCT test - 1 week | 15 (2.9) | 10.8 (2.2)
  activity of an induced HCT test - 2 weeks | 22 (3.1) | 10.4 (3.3)
  activity of an induced HCT test - 6 weeks | 26 (3.4) | 10.9 (3.8)
  percentage of HCT-positive cells - baseline | 7 (3.2) | 6 (2)
  percentage of HCT-positive cells - 1 week | 11 (2.6) | 7.4 (2.3)
  percentage of HCT-positive cells - 2 weeks | 15 (2.9) | 7.2 (1.9)
  percentage of HCT-positive cells - 6 weeks | 17 (3.6) | 6.7 (1.8)

6. Secondary Outcome: Immunophenotype of Blood Lymphocytes in Patients With COPD
Description: Immunophenotype of blood lymphocytes in patients with COPD at baseline, 1, 2 and 6 weeks after PCV13 and PPV23 vaccination. It was pre-specified to report data from only the "COPD - Prevenar-13" and the "COPD - Pneumo-23" Arms/Groups for this Outcome Measure". This is due to the fact that we tried to study the effect of PCV13 and PPV23 on immunity values. The study of the immunological effects of vaccination in the early post-vaccination period was carried out in 2 groups of patients: 20 patients with COPD vaccinated with PCV13; 20 patients with COPD vaccinated with PPV23. These patients were selected from patients of the main groups (COPD - Prevenar-13 (1), COPD - Pneumo-23 (3)).
Time Frame: Baseline, 1, 2, 6 weeks after PCV13 and PPV13 vaccination
Population: CD3+, CD3+CD4+, CD3+CD8+, CD19+, CD3-CD16+CD56+, CD3+CD16+CD56+, CD3-HLA DR+, CD3+HLA DR+
Measure: Mean (Standard Deviation); unit: % of cells
Groups:
- COPD - Prevenar-13 (1): 20 patients with COPD. Prevenar-13 (PCV13) vaccination.
- COPD - Pneumo-23 (3): 20 patients with COPD. Pneumo-23 (PPV23) vaccination.
Arm/Group | COPD - Prevenar-13 (1) | COPD - Pneumo-23 (3)
Number analyzed (Participants) | 20 | 20
% of cells
  CD3+, baseline | 67.3 (4.8) | 69.6 (5.9)
  CD3+, 1 week after vaccination | 69.7 (3.8) | 69.9 (6.9)
  CD3+, 2 weeks after vaccination | 69 (2.8) | 71.3 (5.9)
  CD3+, 6 weeks after vaccination | 66.9 (3.7) | 69.9 (6.1)
  CD3+CD4+, baseline | 35.9 (7.6) | 35.9 (2.2)
  CD3+CD4+, 1 week after vaccination | 40.7 (4.5) | 37.3 (2.7)
  CD3+CD4+, 2 weeks after vaccination | 39.4 (5.8) | 36.9 (2.8)
  CD3+CD4+, 6 weeks after vaccination | 38.9 (5.4) | 37.8 (2.5)
  CD3+CD8+, baseline | 26.2 (6.9) | 26.7 (2.5)
  CD3+CD8+, 1 week after vaccination | 23.5 (3.5) | 26.9 (2.3)
  CD3+CD8+, 2 weeks after vaccination | 32.4 (5.1) | 27.6 (1.9)
  CD3+CD8+, 6 weeks after vaccination | 33.3 (5.2) | 27.9 (1.2)
  CD19+, baseline | 12.5 (3.9) | 13.7 (3.3)
  CD19+, 1 week after vaccination | 13.3 (3) | 15.6 (2.7)
  CD19+, 2 weeks after vaccination | 11 (2.5) | 14.9 (2.9)
  CD19+, 6 weeks after vaccination | 15.1 (3.8) | 14.5 (3.1)
  CD3-CD16+CD56+, baseline | 18.3 (3.9) | 17.3 (2.3)
  CD3-CD16+CD56+, 1 week after vaccination | 14 (3) | 16.6 (2.2)
  CD3-CD16+CD56+, 2 weeks after vaccination | 13 (3.9) | 16.2 (2.2)
  CD3-CD16+CD56+, 6 weeks after vaccination | 16.8 (3.7) | 16.7 (2.2)
  CD3+CD16+CD56+, baseline | 11 (3.8) | 10.6 (2.6)
  CD3+CD16+CD56+, 1 week after vaccination | 11 (4.2) | 11.9 (2.3)
  CD3+CD16+CD56+, 2 weeks after vaccination | 22.5 (7.3) | 11.8 (2.6)
  CD3+CD16+CD56+, 6 weeks after vaccination | 17 (5.3) | 10.8 (2.2)
  CD3-HLA DR+, baseline | 8.6 (4.2) | 10.7 (2.9)
  CD3-HLA DR+, 1 week after vaccination | 13 (3.8) | 11.9 (2.9)
  CD3-HLA DR+, 2 weeks after vaccination | 7 (4.9) | 12.3 (2.4)
  CD3-HLA DR+, 6 weeks after vaccination | 9.5 (5.1) | 11.3 (2.9)
  CD3+HLA DR+, baseline | 12.1 (3.5) | 11.5 (1.9)
  CD3+HLA DR+, 1 week after vaccination | 11.8 (4.2) | 12.5 (1.3)
  CD3+HLA DR+, 2 weeks after vaccination | 10.1 (3.2) | 12.3 (1.5)
  CD3+HLA DR+, 6 weeks after vaccination | 16.2 (4.5) | 11.6 (1.5)

7. Secondary Outcome: IgA, IgM, IgG, IgE, Circulating Immune Complexes (CIC)
Description: IgA, IgM, IgG, IgE, circulating immune complexes (CIC) in serum at baseline, 1, 2 and 6 weeks after vaccination. It was pre-specified to report data from only the "COPD - Prevenar-13" and the "COPD - Pneumo-23" Arms/Groups for this Outcome Measure". This is due to the fact that we tried to study the effect of PCV13 and PPV23 on immunity values. The study of the immunological effects of vaccination in the early post-vaccination period was carried out in 2 groups of patients: 20 patients with COPD vaccinated with PCV13; 20 patients with COPD vaccinated with PPV23. These patients were selected from patients of the main groups (COPD - Prevenar-13 (1), COPD - Pneumo-23 (3)).
Time Frame: Baseline, 1, 2, 6 weeks after PCV13 and PPV13 vaccination in COPD
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | COPD - Prevenar-13 (1) | COPD - Pneumo-23 (3)
Number analyzed (Participants) | 20 | 20
g/l
  IgA, baseline | 3.57 (1.18) | 3.33 (0.55)
  IgA, 1 week after vaccination | 3.74 (1.25) | 3.39 (0.58)
  IgA, 2 weeks after vaccination | 3.79 (1.26) | 3.52 (0.58)
  IgA, 6 weeks after vaccination | 3.63 (1.13) | 3.56 (0.61)
  IgM, baseline | 1 (0.21) | 1.26 (0.47)
  IgM, 1 week after vaccination | 1.25 (0.62) | 1.3 (0.47)
  IgM, 2 weeks after vaccination | 1 (0.17) | 1.3 (0.51)
  IgM, 6 weeks after vaccination | 1 (0.23) | 1.34 (0.49)
  IgG, baseline | 12.8 (1.13) | 11.6 (2.5)
  IgG, 1 week after vaccination | 12.9 (0.8) | 11.7 (2.5)
  IgG, 2 weeks after vaccination | 13.4 (1.04) | 11.9 (2.5)
  IgG, 6 weeks after vaccination | 13.1 (0.57) | 11.8 (2.5)
  IgE, baseline | 120 (42) | 120 (39)
  IgE, 1 week after vaccination | 126 (87) | 118 (42)
  IgE, 2 weeks after vaccination | 118 (74) | 120 (34)
  IgE, 6 weeks after vaccination | 119 (51) | 120 (35)
  CIC, baseline | 0.067 (0.02) | 0.073 (0.01)
  CIC, 1 week after vaccination | 0.086 (0.01) | 0.077 (0.01)
  CIC, 2 weeks after vaccination | 0.079 (0.015) | 0.08 (0.01)
  CIC, 6 weeks after vaccination | 0.073 (0.016) | 0.079 (0.01)

8. Secondary Outcome: CD45RO
Description: CD45RO expression on lymphocytes in serum at baseline, 1 and 4 years after vaccination. These patients were selected from patients of the main groups.
Time Frame: Baseline, 1 and 4 years after vaccination
Measure: Mean (Standard Deviation); unit: U
Groups:
- COPD With Prevenar-13 (1): 32 patients with COPD. Standard therapy with Prevenar-13.
  Prevenar-13: Conjugate 13 serotype pneumococcal vaccine
- Asthma With Prevenar 13 (2): 33 patients with asthma. Standard therapy with Prevenar 13.
  Prevenar-13: Conjugate 13 serotype pneumococcal vaccine
- COPD With Pneumo-23 (3): 23 patients with COPD. Standard therapy with Pneumo-23.
  Pneumo-23: Polysaccharide 23-valent pneumococcal vaccine.
Arm/Group | COPD With Prevenar-13 (1) | Asthma With Prevenar 13 (2) | COPD With Pneumo-23 (3) | Asthma With Pneumo-23 (4) | COPD With Pneumo-23/Prevenar-13 (5) | Asthma With Pneumo-23/Prevenar-13 (6) | COPD With Prevenar-13/Pneumo-23 (7) | Asthma With Prevenar-13/Pneumo-23 (8)
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
U
  CD45RO, baseline | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01)
  CD45RO, 1 year after vaccination | 0.43 (0.04) | 0.2 (0.02) | 0.1 (0.01) | 0.15 (0.01) | 0.47 (0.06) | 0.67 (0.13) | 0.71 (0.12) | 0.73 (0.15)
  CD45RO, 4 years after vaccination | 0.24 (0.03) | 0.2 (0.015) | 0.05 (0.01) | 0.1 (0.01) | 0.31 (0.02) | 0.32 (0.08) | 0.59 (0.1) | 0.59 (0.12)

9. Secondary Outcome: Specific IgG Levels in Vaccinated Patients With COPD to S. Pneumoniae Serotypes
Description: Mean specific IgG levels in vaccinated patients with COPD to S. pneumoniae serotypes at baseline, 6 and 12 months after vaccination
Time Frame: Baseline, 1 and 12 months after vaccination
Measure: Median (Inter-Quartile Range); unit: U/ml
Groups:
- COPD - Prevenar-13: 32 patients with COPD. Prevenar-13 (PCV13) vaccination.
- COPD - Pneumo-23: 23 patients with COPD. Pneumo-23 (PPV23) vaccination.
- COPD - Pneumo-23/Prevenar-13: 32 patients with COPD, PPV23/PCV13.
  PPV23 vaccination was first, PCV13 vaccination was after 12 months after PPV23.
- COPD - Prevenar-13/Pneumo-23: 25 patients with COPD. PCV13/PPV23 vaccination.
  PCV13 vaccination was first, PPV23 vaccination was after 2 months after PCV13.
Arm/Group | COPD - Prevenar-13 | COPD - Pneumo-23 | COPD - Pneumo-23/Prevenar-13 | COPD - Prevenar-13/Pneumo-23
Number analyzed (Participants) | 32 | 23 | 32 | 25
U/ml
  Baseline | 69.7 [40.9 to 113.1] | 66.9 [44 to 92.1] | 87.5 [61.7 to 132.3] | 88 [57.1 to 121.9]
  6 months after vaccination | 132.7 [88.9 to 179.9] | 106.9 [52 to 284.5] | 119.4 [76.9 to 160.9] | 142.2 [90.3 to 200.5]
  12 months after vaccination | 112.9 [69.2 to 157.1] | 94.9 [48 to 253.1] | 0 [0 to 0] | 136 [97.4 to 193.4]

ADVERSE EVENTS:
Time Frame: 7 days after vaccination
Arm/Group | COPD - Prevenar-13 (1) | Asthma - Prevenar-13 (2) | COPD - Pneumo-23 (3) | Asthma - Pneumo-23 (4) | COPD - Pneumo-23/Prevenar-13 (5) | Asthma - Pneumo-23/Prevenar-13 (6) | COPD - Prevenar-13/Pneumo-23 (7) | Asthma - Prevenar-13/Pneumo-23 (8)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/23 | 0/25 | 0/32 | 0/18 | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/23 | 0/25 | 0/32 | 0/18 | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No